CLINICAL TRIAL: NCT04760080
Title: Adjunction of Hydroxychloroquine in Patients With a Metastatic Melanoma Who Are Resistant to BRAF and MEK Inhibitors : a Retrospective Case-control Study.
Brief Title: Association of Hydroxychloroquine, BRAF and MEK Inhibitors in Metastatic Melanoma : a Retrospective Case-control Study.
Acronym: CHLORO-DATRAM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1230
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Dermatology and Oncology
Keywords: metastatic melanoma; BRAF inhibitor; MEK inhibitor; hydroxychloroquine; autophagy
MeSH Terms: conditions — Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a metastatic melanoma treated by dabrafenib/trametinib and hydroxychloroquine.: Patients with a metastatic melanoma treated by dabrafenib/trametinib and hydroxychloroquine after acquired resistance to dabrafenib/trametinib.
  Patients treated
  * for a BRAF mutated metastatic melanoma in Pr Dalle's dermatology ward at Centre Hospitalier Lyon Sud,
  * From January 2008 to June 2020
  * who received a treatment by immunotherapy before receiving a treatment by dabrafenib/trametinib
  * who became resistant to dabrafeib/trametinib
  * and received after disease progression a treatment by dabrafenib/trametinib and hydroxychloroquine
  Interventions: Other: pre-treatment data; Other: during study treatment
- Patients with a metastatic melanoma treated by cytotoxic chemotherapy.: Patients with a metastatic melanoma treated by cytotoxic chemotherapy after acquired resistance to dabrafenib/trametinib.
  Patients treated
  * for a BRAF mutated metastatic melanoma in Pr Dalle's dermatology ward at Centre Hospitalier Lyon Sud,
  * From January 2008 to June 2020
  * who received a treatment by immunotherapy before receiving a treatment by dabrafenib/trametinib
  * who became resistant to dabrafeib/trametinib
  * and received after disease progression under dabrafenib/trametinib a treatment by cytotoxic chemotherapy

INTERVENTIONS:
Other: pre-treatment data — We will evaluate in all patients pre-treatment data :
  * Melanoma staging at treatment initiation
  * Melanoma characteristics at initial diagnosis
  * Number and location of metastasis
  * Performans status
  * Demographic information
  Groups: Patients with a metastatic melanoma treated by dabrafenib/trametinib and hydroxychloroquine.
Other: during study treatment — We will evaluate in all patients during study treatment :
  * Rate of adverse events
  * Type of adverse events
  * Radiological response to treatment by CTscans that are routinely performed every three months.
  Groups: Patients with a metastatic melanoma treated by dabrafenib/trametinib and hydroxychloroquine.

SUMMARY:
Patients with a BRAF mutated melanoma are usually treated in France by a first line of immunotherapy followed by a second line that combines a BRAF inhibitor (dabrafenib, vemurafenib, encorafenib) and a MEK inhibitor (trametinib, cobimetinib, binimetinib).

The combination dabrafenib/trametinib is initially very efficient but it is unfortunately limited because acquired resistances usually occur after a year of treatment. Patients who become resistant to dabrafenib/trametinib and immunotherapy, unfortunately do not have an approved effective treatment at their disposal. They usually receive a palliative chemotherapy by dacarbazine or fotemustine, and they have a mean overall survival that is less than three months.

Activation of autophagy in presence of BRAF and MEK inhibitors is a known mechanism of resistance to BRAF/MEK inhibitors. Hydroxychloroquine is an autophagy inhibitor and it has been suggested in vitro that it could decrease resistance to BRAF/MEK inhibitors.

Following the positive results in 2018 of a phase I/II study in the USA that showed the efficacy and the absence of toxicity of the association of Dabrafenib, Trametinib and hydroxychloroquine when used as a first line treatement, we proposed to our patients who had become resistant to the dabrafenib/trametinib combination, to pursue their treatment beyond progression and to receive in addition hydroxychloroquine.

This prescription was initiated in patients for whom no further therapeutic options were available, after validation by a multidisciplinary tumor board. All patients were informed that the combination dabrafenib/trametinib/hydroxychloroquine was not approved by a regulatory agency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic melanoma with an activating BRAF mutation
* Who received at least one line of immunotherapy
* Whose disease is resistant to a BRAF inhibitor used as a single agent or in combination with a MEK inhibitor
* Who received either cytotoxic chemotherapy or the combination dabrafenib + trametinib + hydroxychloroquine after disease progression to dabrafenib/trametinib from January 2008 to June 2020 in the Dermatology ward of the Lyon Sud Hospital

Exclusion Criteria:

* Patients who did not received an immunotherapy prior to dabrafenib/trametinib treatment
* Absence of tumor board validation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated
  * for a BRAF mutated metastatic melanoma in Pr Dalle's dermatology ward at Centre Hospitalier Lyon Sud,
  * From January 2008 to June 2020
  * who received a treatment by immunotherapy before receiving a treatment by dabrafenib/trametinib
  * who became resistant to dabrafeib/trametinib
  * and received after disease progression either a treatment by dabrafenib/trametinib and hydroxychloroquine or a cytotoxic chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of progression free survival (PFS) in patients who are resistant to dabrafenib/trametinib who receive dabrafenib/trametinib/hydroxychloroquine despite tumor progression versus cytotoxic chemotherapy | Patients treated from January 2008 to June 2020 will be included retrospectively in this study. Data cut off will be defined in June 2020.
  Progression Free Survival: the length of time during and after the treatment of a cancer, that a patient lives with the disease but it does not get worse

CONTACTS AND LOCATIONS:
Overall Officials: Victoire REYNAUD, MD, Principal Investigator — Centre Hospitalier Lyon Sud, Dermatology unit
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France